CLINICAL TRIAL: NCT06622408
Title: Contribution of Virtual Reality in the Management of Patients Undergoing Scheduled Cesarean Section - VR-SCS Study (Virtual Reality and Schedulded Cesarean Section)
Brief Title: Contribution of Virtual Reality in the Management of Patients Undergoing Scheduled Cesarean Section - VR-SCS
Acronym: VR-SCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-AOIP-05
Record Dates: First submitted 2024-07-18; First posted 2024-10-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Women's Health; Perinatal Care; Cesarean; Analgesia
Keywords: cesarean; analgesia; women
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scheduled caesarean delivery (Experimental): Use of virtual reality headset during patient admission to the OR for cesarean section.
  Interventions: Other: HypnoVR© virtual reality headset

INTERVENTIONS:
Other: HypnoVR© virtual reality headset — Adherence to the use of the virtual reality headset will be reported by a percentage of use at each stage of care.

SUMMARY:
Cesarean deliveries account for 20.7% of all deliveries in France, according to the latest perinatal survey. At Nice University Hospital, the C-section rate over the last 5 years is around 19%.

Caesarean section patients are at greater risk of developing symptoms of anxiety, stress and depression. The post-operative period is also more painful, and there is a positive correlation between immediate post-operative pain and the risk of developing chronic pelvic pain. Numerous attempts to reduce these symptoms have been evaluated, including music therapy, relaxation techniques, acupressure and the use of preoperative melatonin.

Virtual reality has demonstrated its effectiveness in reducing pain and anxiety in other disciplines, notably pediatric surgery and neurosurgery.

In particular, several trials have demonstrated a reduction in anxiety in the paediatric population and, for pelvic procedures under local anaesthetic, during prostate biopsies or hysteroscopy in consultation, with a reduction in anxiety and pain respectively.

It has been used to provide information by showing a film about the caesarean section procedure, and has been shown to be effective in terms of patient satisfaction, but without being able to demonstrate a significant reduction in anxiety (p=0.06).

The use of virtual reality during the entire peri- and intra-operative management process (maternity stay, patient transfer to the operating room, locoregional anesthesia procedure and during the operation) has not been studied in the context of cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Major woman ;
* Female volunteer ;
* Social security affiliation;
* Admitted for scheduled caesarean section with history of caesarean section and patient's refusal to attempt vaginal delivery;
* Informed patients who have signed the informed consent form.

Exclusion Criteria:

* Speaks a language other than French;
* Unbalanced epilepsy;
* People unable to understand (language barrier, cognitive difficulties, cerebral palsy, etc.) and/or apply dietary advice (people institutionalized in nursing homes, retirement homes, prisons, etc.);
* Women claiming to have had a very bad experience during their previous caesarean section.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of a pathway involving the use of virtual reality from patient admission to the cesarean section. | 18 months
  Rate of acceptance of the use of the virtual reality headset during each stage of care (on admission to the maternity ward, in the delivery room before transfer to the operating room, at the patient's request in the caesarean section room after birth (in the absence of skin-to-skin contact with the newborn).

SECONDARY OUTCOMES:
Assessing patients' pain throughout the treatment process | 18 months
  The patient's pain will be assessed according to a VAS from 0 to 100.
Evaluate patient anxiety throughout treatment | 18 months
  The patient's anxiety will be assessed using a VAS from 0 to 100.
Evaluate patient satisfaction throughout the care process | 18 months
  Patient satisfaction will be assessed according to 2 closed questions: "Would you recommend this service to someone close to you? "If you were to have another caesarean section, would you want this care again?
Evaluation of the impact on the course of surgery and the post-operative period | 18 months
  The impact on the course of surgery and the post-operative period will be assessed by Total operative time (in minutes).
Evaluation of the impact on the course of surgery and the post-operative period | 18 months
  The impact on the course of surgery and the post-operative period will be assessed by Amount of blood loss (in mL).
Evaluation of the impact on the course of surgery and the post-operative period | 18 months
  The impact on the course of surgery and the post-operative period will be assessed by the occurrence of nausea/vomiting during the operation.
Evaluation of the impact on the course of surgery and the post-operative period | 18 months
  The impact on the course of surgery and the post-operative period will be assessed by the time between the end of the caesarean section and the patient's first rising (in hours).
Evaluation of the impact on the course of surgery and the post-operative period | 18 months
  The impact on the course of surgery and the post-operative period will be assessed by Time from end of caesarean section to first micturition (in hours).
Assessing the impact on newborns by APGAR | 18 months
  The newborn's condition at birth will be assessed by APGAR at 1 minute of life.
Assessing the impact on newborns by APGAR | 18 months
  The newborn's condition at birth will be assessed by APGAR at 5 minutes of life.
Assessing the impact on newborns by APGAR | 18 months
  The newborn's condition at birth will be assessed by APGAR at 10 minutes of life.
Assessing the impact on newborns | 18 months
  The newborn's condition at birth will be assessed by pH at the cord.
Assessing the impact on newborns | 18 months
  The newborn's condition at birth will be assessed by lactates at the cord (in mmol/L).
Evaluation of the medical team's satisfaction after surgery | 18 months
  The surgeon's satisfaction based on a VAS from 0 to 100 at the end of the procedure and the anesthetist's satisfaction based on a VAS from 0 to 100 at the end of the procedure.
Assessment feasibility | 18 months
  Completion rate of evaluation questionnaires
Evaluation of study refusals | 18 months
  Refusal rate and Reason for refusal to participate (if patient wishes to justify refusal)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nice - Hôpital de l'Archet 2, Nice, Alpes-Maritimes, France